CLINICAL TRIAL: NCT04193436
Title: A PHASE 1, NON-RANDOMIZED, OPEN-LABEL, SINGLE-DOSE, PARALLEL-COHORT STUDY TO COMPARE THE PHARMACOKINETICS OF PF-06835919 IN ADULT PARTICIPANTS WITH VARYING DEGREES OF HEPATIC IMPAIRMENT RELATIVE TO PARTICIPANTS WITHOUT HEPATIC IMPAIRMENT
Brief Title: A STUDY TO COMPARE THE PHARMACOKINETICS OF PF-06835919 IN PARTICIPANTS WITH AND WITHOUT HEPATIC IMPAIRMENT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C1061013; HEPATIC IMPAIRMENT (Other: Alias Study Number); 2019-003480-21 (EudraCT Number)
Record Dates: First submitted 2019-11-11; First posted 2019-12-10 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-06

CONDITIONS: Hepatic Impairment; Healthy Participants
Keywords: Non-alcoholic Fatty Liver Disease; Non-alcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — PF-06835919

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PF-06835919 with severe hepatic impairement (Experimental): This arm includes participants with severe hepatic impairment who will receive a 25mg oral dose of PF-06835919
  Interventions: Drug: PF-06835919 25 mg
- PF-06835919 with moderate hepatic impairement (Experimental): This arm includes participants with moderate hepatic impairment who will receive a 25mg oral dose of PF-06835919
  Interventions: Drug: PF-06835919 25 mg
- PF-06835919 with mild hepatic impairement (Experimental): This arm includes participants with mild hepatic impairment who will receive a 25mg oral dose of PF-06835919
  Interventions: Drug: PF-06835919 25 mg
- PF-06835919 without hepatic impairment (Experimental): This arm includes participants without hepatic impairment who will receive a 25mg oral dose of PF-06835919
  Interventions: Drug: PF-06835919 25 mg

INTERVENTIONS:
Drug: PF-06835919 25 mg — PF-06835919 in 25 mg oral tablet will be administered on Day 1

SUMMARY:
The study is proposed to characterize the effect of varying degrees of hepatic impairment on the plasma PK of PF-06835919

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between the ages of 18 (or the minimum country specific age of consent if >18) and 70 years, inclusive, at the Screening visit:
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Body mass index (BMI) of 17.5 to 35.4 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, ileal resection).

(Participants who have undergone cholecystectomy and/or appendectomy are eligible for this study as long as the surgery occurred more than 6 months prior to Screening)..

* At Screening, participants with a positive result for human immunodeficiency virus (HIV) antibodies, as assessed by sponsor identified central laboratory, with a single repeat permitted to assess eligibility, if needed.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behaviour or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Use of prior/concomitant therapies.
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product used in this study (whichever is longer).
* Participants with known prior participation (ie, randomized and received at least 1 dose of investigational product) in a study involving PF 06835919.
* A positive urine drug test, for illicit drugs, and/or a positive breath alcohol test at Screening. However, participants who have been medially prescribed opiates/opiods or benzodiazepines and report the use of these drugs to the investigator at the screening visit will be allowed to participate.
* Male participants with partners who are currently pregnant.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing and until the follow-up contact.
* History of sensitivity to heparin or heparin induced thrombocytopenia, only if heparin is used to flush intravenous catheters used during serial blood collections.
* Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of the protocol.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium
- Pharmaceutical Research Associates CZ, s.r.o., Prague, Czechia
- Summit Clinical Research, s.r.o.,, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1061013

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 34 participants were screened, of whom 11 had screen failure and 23 entered the study. There were 6, 6, 6 and 5 participants in the without hepatic impairment group, mild hepatic impairment group, moderate hepatic impairment group and severe hepatic impairment group, respectively. All of the 23 treated participants received their assigned treatment, and no participant discontinued.
Groups:
- Without Hepatic Impairment: This arm included participants without hepatic impairment who received a 25 mg single oral dose of PF-06835919 on Day 1.
- Mild Hepatic Impairment: This arm included participants with mild hepatic impairment who received a 25 mg single oral dose of PF-06835919 on Day 1.
- Moderate Hepatic Impairment: This arm included participants with moderate hepatic impairment who received a 25 mg single oral dose of PF-06835919 on Day 1.
- Severe Hepatic Impairment: This arm included participants with severe hepatic impairment who received a 25 mg single oral dose of PF-06835919 on Day 1.
Period: Overall Study
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Started | 6 | 6 | 6 | 5
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants randomly assigned to investigational product and who took at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Total
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 23
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 64 years (inclusive) | 2 | 4 | 3 | 2 | 11
  ≥65 years | 4 | 2 | 3 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 0 | 7
  Male | 2 | 4 | 5 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 5 | 5 | 22
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 5 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinite Time (AUCinf) of PF-06835919
Description: AUCinf was defined as area under the plasma concentration time curve from time 0 extrapolated to infinite time.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 ,72, 96 ,120 hours post dose on Day 1.
Population: The PK parameter analysis population was defined as all participants dosed who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 5
nanogram*hour per milliliter (ng*hr/mL) | 14090 (29) | 13090 (36) | 18930 (34) | 19630 (28)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; The effect of the hepatic impairment on PK parameter AUCinf were assessed by constructing 90% confidence intervals around the estimated difference between each of the Test (impaired) cohorts and the Reference (without hepatic impairment) cohort using a one-way analysis of variance (ANOVA) model based on natural log transformed data; Test type: Other; Ratio (%) of Adjusted Means = 92.89, 90% CI 2-sided [68.15 to 126.60]
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; The effect of the hepatic impairment on PK parameter AUCinf were assessed by constructing 90% confidence intervals around the estimated difference between each of the Test (impaired) cohorts and the Reference (without hepatic impairment) cohort using a one-way ANOVA model based on natural log transformed data; Test type: Other; Ratio (%) of Adjusted Means = 134.40, 90% CI 2-sided [98.61 to 183.17]
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio (%) of Adjusted Means = 139.33, 90% CI 2-sided [100.69 to 192.78]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of PF-06835919
Description: Cmax was defined as maximum plasma concentration of PF-06835919 and observed directly from data.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 ,72, 96 ,120 hours post dose on Day 1.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 5
ng/mL | 1310 (17) | 1143 (47) | 1340 (28) | 1098 (31)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; The effect of the hepatic impairment on PK parameter Cmax were assessed by constructing 90% confidence intervals around the estimated difference between each of the Test (impaired) cohorts and the Reference (without hepatic impairment) cohort using a one-way ANOVA model based on natural log transformed data; Test type: Other; Ratio (%) of Adjusted Means = 87.20, 90% CI 2-sided [63.61 to 119.53]
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio (%) of Adjusted Means = 102.24, 90% CI 2-sided [74.59 to 140.15]
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio (%) of Adjusted Means = 83.78, 90% CI 2-sided [60.18 to 116.62]

3. Primary Outcome: Unbound Area Under The Plasma Concentration-Time Curve From Time 0 Extrapolated To Infinite Time (AUCinf,u) of PF-06835919
Description: AUCinf,u was defined as unbound area under the plasma concentration time curve from time 0 extrapolated to infinite time.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 ,72, 96 ,120 hours post dose on Day 1.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 5
ng*hr/mL | 612.6 (29) | 746.2 (22) | 1093 (43) | 1199 (34)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; The effect of the hepatic impairment on PK parameter AUCinf,u were assessed by constructing 90% confidence intervals around the estimated difference between each of the Test (impaired) cohorts and the Reference (without hepatic impairment) cohort using a one-way ANOVA model based on natural log transformed data; Test type: Other; Ratio (%) of Adjusted Means = 121.81, 90% CI 2-sided [88.69 to 167.31]
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio (%) of Adjusted Means = 178.50, 90% CI 2-sided [129.96 to 245.18]
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio (%) of Adjusted Means = 195.73, 90% CI 2-sided [140.31 to 273.03]

4. Primary Outcome: Unbound Maximum Plasma Concentration (Cmax,u) of PF-06835919
Description: Cmax,u was defined as unbound maximum plasma concentration.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 ,72, 96 ,120 hours post dose on Day 1.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 5
ng/mL | 56.93 (18) | 65.16 (32) | 77.45 (26) | 67.10 (30)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; The effect of the hepatic impairment on PK parameter Cmax,u were assessed by constructing 90% confidence intervals around the estimated difference between each of the Test (impaired) cohorts and the Reference (without hepatic impairment) cohort using a one-way ANOVA model based on natural log transformed data; Test type: Other; Ratio (%) of Adjusted Means = 114.45, 90% CI 2-sided [88.13 to 148.63]
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio (%) of Adjusted Means = 136.04, 90% CI 2-sided [104.75 to 176.67]
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio (%) of Adjusted Means = 117.87, 90% CI 2-sided [89.61 to 155.03]

5. Primary Outcome: Fraction of Drug Unbound (fu) of PF-06835919
Description: The fraction of PF-06835919 unbound in plasma (fu) was determined at approximately the expected Tmax in each participant.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 ,72, 96 ,120 hours post dose on Day 1.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 5
ratio | 0.04345 (5) | 0.05704 (21) | 0.05780 (18) | 0.06111 (14)

6. Secondary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An serious adverse event (SAE) was defined as an AE: 1. resulting in death, 2. was life-threatening, 3. required inpatient hospitalization or prolongation of existing hospitalization, 4. resulted in persistent disability, 5. was a congenital anomaly/birth defect, or considered to be an important medical event. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent AE (TEAE) was defined as an AE with onset date occurring during the on-treatment period. AEs included all SAEs and non-SAEs.
Time Frame: Baseline (Day 1) up to follow-up (Day 31)
Population: The safety analysis population was defined as all participants randomly assigned to investigational product and who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 5
Participants
  With all-causality TEAE | 0 | 0 | 1 | 1
  With treatment-related TEAE | 0 | 0 | 1 | 0
  With SAE | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Change (Chg) From Baseline in Laboratory Tests
Description: To determine if there were any clinically significant laboratory abnormalities, hematology (hemoglobin, hematocrit, erythrocytes, mean corpuscular hemoglobin, mean corpuscular volume, platelet count, lymphocytes, neutrophils, activated partial thromboplastin time, prothrombin time, prothrombin intl. normalized ratio), clinical chemistry (bilirubin, direct and indirect bilirubin, gamma glutamyl transferase, albumin, urea nitrogen, glucose) and urinalysis (glucose, protein, hemoglobin, urobilinogen, nitrite) tests were assessed. Each parameter was evaluated against commonly used and widely accepted criteria.
Time Frame: Baseline (Day 1) up to Day 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 5
Participants
  Hemoglobin (g/dL) <0.8*lower limit of normal (LLN): number analyzed (Participants) | 6 | 6 | 6 | 4
  Hemoglobin (g/dL) <0.8*lower limit of normal (LLN) | 0 | 0 | 1 | 0
  Hematocrit (%) <0.8*LLN: number analyzed (Participants) | 6 | 6 | 6 | 4
  Hematocrit (%) <0.8*LLN | 0 | 0 | 1 | 0
  Erythrocytes (10^6/mm3) <0.8*LLN: number analyzed (Participants) | 6 | 6 | 6 | 4
  Erythrocytes (10^6/mm3) <0.8*LLN | 0 | 0 | 1 | 2
  Ery. Mean Corpuscular Volume (um^3) >1.1*upper limit of normal (ULN): number analyzed (Participants) | 6 | 6 | 6 | 4
  Ery. Mean Corpuscular Volume (um^3) >1.1*upper limit of normal (ULN) | 0 | 0 | 1 | 1
  Ery. Mean Corpuscular Hemoglobin (pg/cell) >1.1*ULN: number analyzed (Participants) | 6 | 6 | 6 | 4
  Ery. Mean Corpuscular Hemoglobin (pg/cell) >1.1*ULN | 0 | 0 | 0 | 1
  Platelets (10^3/mm3) <0.8*LLN: number analyzed (Participants) | 6 | 6 | 6 | 4
  Platelets (10^3/mm3) <0.8*LLN | 0 | 0 | 3 | 4
  Lymphocytes (10^3/mm3) <0.8*LLN: number analyzed (Participants) | 6 | 6 | 6 | 4
  Lymphocytes (10^3/mm3) <0.8*LLN | 0 | 0 | 1 | 0
  Neutrophils (10^3/mm3) <0.8*LLN: number analyzed (Participants) | 6 | 6 | 6 | 4
  Neutrophils (10^3/mm3) <0.8*LLN | 0 | 0 | 0 | 1
  Activated Partial Thromboplastin Time (sec) >1.1*ULN | 0 | 0 | 1 | 2
  Prothrombin Time (sec) >1.1*ULN | 0 | 0 | 5 | 5
  Prothrombin Intl. Normalized Ratio >1.1*ULN | 0 | 0 | 5 | 5
  Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 1 | 5
  Direct Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 4 | 5
  Indirect Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 0 | 2
  Gamma Glutamyl Transferase (U/L) >3.0*ULN | 0 | 0 | 2 | 0
  Albumin (g/dL) <0.8*LLN | 0 | 0 | 0 | 1
  Urea Nitrogen (mg/dL) >1.3*ULN | 0 | 1 | 0 | 0
  Glucose (mg/dL) >1.5*ULN | 0 | 1 | 1 | 0
  URINE Glucose (mg/dL) ≥1 | 0 | 1 | 0 | 0
  URINE Protein (mg/dL) ≥1 | 0 | 0 | 0 | 1
  URINE Hemoglobin ≥1 | 0 | 0 | 1 | 1
  Urobilinogen (EU/dL) ≥1 | 0 | 0 | 0 | 5
  Nitrite ≥1 | 1 | 0 | 0 | 1

8. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-Lead Electrocardiograms (ECGs)
Description: ECG endpoints (PR interval, QRS interval, QT interval and QTcF) meeting the criteria of potential clinical concern were summarized by treatment using categories as defined: 1. PR max. ≥300ms, %Chg ≥25/50%; 3. QRS max. ≥140ms，%Chg ≥50%; 3.maximum post-dose QTcF 450 - ≤480msec, 480 - ≤500msec and >500msec, 30<Chg≤60 and Chg>60.
Time Frame: Baseline (Day 1) up to Day 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 5
Participants
  PR Interval Value ≥300 msec | 0 | 0 | 0 | 0
  PR Interval %Chg ≥25/50% | 0 | 0 | 0 | 0
  QRS Interval Value ≥140 msec | 0 | 0 | 0 | 0
  QRS Interval %Chg ≥50% | 0 | 0 | 0 | 0
  QT Interval Value >500 msec | 0 | 0 | 0 | 1
  QTcF (msec) 450< Value ≤480 | 0 | 0 | 0 | 2
  QTcF (msec) 480< Value ≤500 | 0 | 0 | 0 | 1
  QTcF (msec) Value >500 | 0 | 0 | 0 | 0
  QTcF (msec) 30< Chg ≤60 | 0 | 0 | 1 | 0
  QTcF (msec) Chg >60 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to follow-up (Day 31)
Description: All participants randomly assigned to investigational product and who took at least 1 dose of investigational product.
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Without Hepatic Impairment (N=6) | Mild Hepatic Impairment (N=6) | Moderate Hepatic Impairment (N=6) | Severe Hepatic Impairment (N=5)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT04193436/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT04193436/SAP_001.pdf